CLINICAL TRIAL: NCT04738253
Title: Study on Post-stroke Patients With Limited Range of Motion in the Shoulder Joint Whose Ultrasonographic Findings Show Adhesive Capsulitis and Its Associated Clinical Factors.
Brief Title: Correlation Between Ultrasonography Finding and Shoulder Range of Motion in Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yeungnam University Hospital (Other)
Responsible Party: Principal Investigator, Dong Gyu Lee, Assistant professor, Yeungnam University Hospital
Other Study IDs: 2020-10-015-002
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Stroke; Frozen Shoulder
Keywords: Cerebral Stroke; Frozen Shoulder; ultrasonography
MeSH Terms: conditions — Stroke; Bursitis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Stroke patients with limitation of range of motion on the affected shoulder.
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — The ultrasound measurement s of the axillary recess capsule thickness.

SUMMARY:
Limitation of range of motion in the shoulder joints is common in stroke patients. The causes are stiffness, CRPS, and frozen shoulder. The purpose of this study was to investigate the relationship between frozen shoulder and shoulder LOM in patients with cerebral infarction using ultrasonography.

DETAILED DESCRIPTION:
Ultrasound examination was performed on 50 patients with limited range of motion of the shoulder joint among inpatients or outpatients in the Department of Rehabilitation Medicine of our hospital, who had a stroke of fewer than 2 years, and the findings suitable for adhesive capsulitis, namely the thickness of the joint capsule in the axillary concave Identify those with thickened findings. Their shoulder power rating, passive range of motion, stiffness evaluation (Modified Ashworth Scale, MAS), and the presence or absence of Reflex Sympathetic Dystrophy (RSD) were evaluated, and the relationship with ultrasound findings was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Those who have been diagnosed with a stroke through CT or MRI within the last 2 years
* Those who are over 19 years old
* Those who have limitations in the range of motion of the shoulder joint

Exclusion Criteria:

* Those diagnosed with adhesive arthritis prior to the onset of stroke
* Patients with a severe shoulder trauma
* Those who performed shoulder surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the cerebral stroke patients with limitation of range of motion on affected shoulder.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Range of motion of shoulder joint | day 1
  A goniometer is an instrument which measures the available range of motion at a joint.Flexion, Extension,Adduction,Abduction, Internal Rotation,External rotation

SECONDARY OUTCOMES:
MAS(Modified Ashworth Scale) of elbow Flexor | day 1
  The Modified Ashworth Scale is a well known and commonly used scale in clinical trials with spasticity. It was considered to be the best clinical tool for measuring resistance to movement. It was used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).

CONTACTS AND LOCATIONS:
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided